CLINICAL TRIAL: NCT05025670
Title: Tracking Response in Advance of Investigational Trials, Borderline Study
Acronym: TRAIT-BOR
Status: Completed | Type: Observational
Sponsor: Adams Clinical (Network)
Responsible Party: Sponsor
Other Study IDs: TRAIT-BOR-101
Record Dates: First submitted 2021-08-20; First posted 2021-08-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Supportive psychotherapy — Participants will receive monthly 30-45 minute supportive psychotherapy sessions. Supportive psychotherapy is an integrative and eclectic psychotherapeutic approach, based upon the individual's needs and symptoms. It draws from elements of a variety of psychotherapeutic disciplines, including cognitive-behavior, psychodynamic, and interpersonal therapies.

SUMMARY:
TRAIT-BOR is an open-label psychotherapy treatment study for adults who meet the diagnostic criteria for Borderline Personality Disorder (BPD) and are seeking enrollment in a clinical trial of a novel compound to treat BPD. The current study seeks to determine if there are therapeutic benefits to more infrequent, short term, or longer term supportive psychotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Participant has signed an ICF prior to any study-specific procedures being performed.
* Participant has a diagnosis of Borderline Personality Disorder, per DSM-5 criteria, as confirmed on the MINI, and ≥ 16 AAPI-CR total score.
* Participant is in good physical health, and, in the opinion of the investigator, is a suitable candidate for treatment with monthly supportive psychotherapy.
* Participant is 18 to 65 years old.
* For participants already receiving psychotherapy, including Dialectical Behavioral Therapy (DBT), they must continue their regular course of treatment for the duration of the current study.

Exclusion Criteria:

* Participant is pregnant, breast-feeding, or planning to become pregnant.
* A history or presence of a clinically significant hepatic, renal, gastrointestinal, cardiovascular, endocrine, respiratory, immunologic, hematologic, dermatologic, or neurologic abnormality, which in the opinion of the investigator may impact participant safety or study results.
* Participant has a history of any psychiatric condition other than BPD, which in the opinion of the investigator is primary, or any other psychiatric or neurologic disorder or symptom that could pose undue risk to the participant or compromise the study.
* Any participant who represents an acute suicidal risk in the opinion of the investigator, as defined by a "yes" response to suicidal ideation on questions 4 or 5, or answer "yes" to suicidal behavior questions on the CSSR-S within 90 days of screening.
* Any participant who represents an acute homicidal risk in the opinion of the investigator.
* Moderate or severe substance use disorder within 90 days prior to screen, according to DSM-5 criteria that in the opinion of the investigator could pose undue risk to the participant, or compromise the study.
* Any condition that, in the opinion of the investigator, makes the participant unsuitable for the study.
* Participants who require ongoing treatment with typical antipsychotics.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 to 65 years old, who meet criteria for BPD, and who have expressed interest in participating in a clinical trial of an investigational product for treatment of BPD.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Stability of symptoms and treatment response as defined as change in total scores on the Agitation-Aggression Psychiatric Inventory - Clinician Report (AAPI-CR) from Baseline/Day 0 to End of Cycle (EOC)/Day 90. | 90 days
  Total scores on the AAPI-CR range from 11 to 275, with higher scores indicating higher levels of agitation and aggression.
Stability of symptoms and treatment response as defined as change in total scores on the self-report Borderline Personality Disorder Checklist (BPDCL) from Baseline/Day 0 to End of Cycle (EOC)/Day 90. | 90 days
  Total scores on the BPDCL range from 47 to 235, with higher scores indicating greater symptom severity.
The proportion of participants who have clinically significant agitation and aggression symptoms, as defined as AAPI-CR Agitation and Aggression (A/A) subscale score ≥ 16 and sum of the A/A subscale severity scores ≥ 6. | Up to 52 weeks

SECONDARY OUTCOMES:
Stability of symptoms and treatment response as defined as change in total score on the Zanarini Rating Scale for Borderline Personality Disorder (ZAN-BPD) from Baseline/Day 0 to End of Cycle (EOC)/Day 90. | 90 days
  Total scores on the ZAN-BPD range from 0 to 36, with higher scores indicating greater symptom severity.
Stability of symptoms and treatment response as defined as change in total scores on the AAPI-CR from Baseline/Day 0 to End of Study (EOS)/Day 224. | Up to 52 weeks
Stability of symptoms and treatment response as defined as change in total scores on the BPDCL from Baseline/Day 0 to End of Study (EOS)/Day 224. | Up to 52 weeks
The proportion of participants who fail to reach response to a brief course of monthly supportive psychotherapy treatment after 3 months. | 90 days
  Defined as either AAPI-CR Total score ≥ 16 by EOC/Day 90 or < 25% decrease in AAPI-CR Total Score from Baseline/Day 0 to EOC/Day 90 and verified by clinician-rated assessment as indicated by a CGI ≥ 4 at EOC/Day 90.
The proportion of participants who fail to reach response to longer term monthly supportive psychotherapy treatment after 8 months. | Up to 52 weeks
  Defined as either AAPI-CR Total score ≥ 16 by EOS/Day 224 or < 25% decrease in AAPI-CR Total Score from Baseline/Day 0 to EOS/Day 224 and verified by clinician-rated assessment as indicated by a CGI ≥ 4 at EOS/Day 224.
The proportion of participants who show a partial response to monthly brief or longer term supportive psychotherapy treatment. | Up to 52 weeks
  Defined as ≥ 25% to < 50% reduction in AAPI-CR Total Score from Baseline/Day 0 to EOC/Day 90 and ≥ 25% to < 50% reduction in AAPI-CR Total Score from Baseline/Day 0 to EOS/Day 224.
The proportion of participants who show a clinically significant response to brief monthly supportive psychotherapy treatment. | 90 days
  Defined as ≥ 50% reduction in AAPI-CR Total Score from Baseline/Day 0 to EOC/Day 90 and verified by clinician-rated assessment as indicated by a CGI ≤ 3 at EOC/Day 90.
The proportion of participants who show a clinically significant response to longer term monthly supportive psychotherapy treatment. | Up to 52 weeks
  Defined as ≥ 50% reduction in AAPI-CR Total Score from Baseline/Day 0 to EOS/Day 224 and verified by clinician-rated assessment as indicated by a CGI ≤ 3 at EOS/Day 224.

OTHER OUTCOMES:
The initial prevalence of comorbid psychiatric symptoms as assessed by the Mini-International Neuropsychiatric Inventory (MINI). | Up to 52 weeks
The proportion of participants who elect to add psychopharmacologic treatment to their monthly supportive psychotherapy by enrolling in an industry-sponsored clinical trial for BPD at the site. | Up to 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Adams Clinical, Watertown, Massachusetts, United States